CLINICAL TRIAL: NCT04320823
Title: Prospective, Randomized, Controlled, Multicenter Clinical Trial to Demonstrate the Safety and Effectiveness of the NexSys® PCS Plasma Collection System With the Percent Plasma Nomogram (PPN) Feature
Brief Title: IMPACT (Improving Plasma Collection) Clinical Trial
Acronym: IMPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haemonetics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: TP-CLN-100467
Record Dates: First submitted 2020-01-03; First posted 2020-03-25 (Actual); Results first posted 2021-04-09 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-03

CONDITIONS: Apheresis Related Hypotension
Keywords: Plasmapheresis (Source plasma collection)

STUDY DESIGN:
Intervention Model Description: Two-arm, randomized, controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Experimental Group (Experimental): Plasma collection using a modified version (version 1.3.90) of NexSys PCS embedded software installed on current FDA-cleared NexSys PCS device hardware (PCS-300-US), with the new plasma collection feature enabled.
  Interventions: Device: Updated Plasma Collection Feature
- Control Group (Active Comparator): Plasma collection using a modified version (version 1.3.90) of NexSys® PCS embedded software installed on current FDA-cleared NexSy PCS device hardware (PCS-300-US), with the new plasma collection feature disabled.
  Interventions: Device: Current Plasma Collection Approach

INTERVENTIONS:
Device: Updated Plasma Collection Feature — Plasma collection using a novel, patented system that supports a more individualized collection approach.
  Arms: Experimental Group
Device: Current Plasma Collection Approach — Plasma collection using the current collection approach.
  Arms: Control Group

SUMMARY:
Prospective, multi-center, randomized, controlled clinical trial to study the safety and effectiveness of a novel plasma collection system software.

DETAILED DESCRIPTION:
Prospective, multi-center, randomized, controlled clinical trial that will be conducted at three source plasma collection centers throughout the United States. The objective of the trial is to study the safety and effectiveness of a novel plasma collection nomogram run on the bi-directionally integrated Haemonetics NexSys PCS® and Haemonetics NexLynk DMS® plasma collection system. Subjects will be randomized into an intervention and control arm. The control arm will donate plasma using the current software. The intervention arm will donate plasma using a novel software that supports a more individualized collection approach.

ELIGIBILITY:
Inclusion Criteria:

* Donors must be qualified to donate plasma per individual site's screening procedures which are in compliance with IQPP standards. If donors do not meet inclusion criteria at subsequent donations but have already been enrolled in the clinical trial, they are eligible to remain in the clinical trial and to donate plasma within the clinical trial once they meet eligibility criteria again, except if they fulfill any of the exclusion criteria listed below.

Exclusion Criteria:

* All subjects meeting any of the exclusion criteria listed below will be permanently excluded from the clinical trial.

  * Subject not able or willing to give consent to participate in the clinical trial.
  * Subject donated plasma outside of the present clinical trial after enrolling in this clinical trial.
  * Subjects are withdrawn from the clinical trial due to safety concerns by the qualified healthcare providers.
  * In addition, all donors for whom a BMI for use in the PPN feature cannot be reliably calculated will be excluded

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Donors must indicate their biological gender.
Enrollment: 3443 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2020-03-27 (Actual); Study Completion 2020-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan F Leitman, MD, Principal Investigator — National Institutes of Health (NIH)
Locations (3):
- United States (3):
  - Octapharma Plasma, Wichita, Kansas
  - Octapharma Plasma, Charlotte, North Carolina
  - Octapharma Plasma, Spokane, Washington

REFERENCES:
- [Derived] Hartmann J, Ragusa MJ, Burchardt ER, Manukyan Z, Popovsky MA, Leitman SF. Personalized collection of plasma from healthy donors: A randomized controlled trial of a novel technology-enabled nomogram. Transfusion. 2021 Jun;61(6):1789-1798. doi: 10.1111/trf.16389. Epub 2021 Apr 21. PMID 33760230

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental Group | Control Group
Started | 1717 | 1726
Completed | 1717 (Includes 47 donors who withdrew from the study after one or more donations.) | 1726 (Includes 38 donors who withdrew from the study after one or more donations.)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Units Other Than Participants: Donations
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Group | Control Group | Total
Number analyzed (Participants) | 1717 | 1726 | 3443
Number analyzed (Donations) | 11362 | 11775 | 23137
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.5 (11.69) | 35.4 (11.10) | 35.4 (11.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 605 | 601 | 1206
  Male | 1112 | 1125 | 2237
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0
    (all) |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 1717 | 1726 | 3443
BMI [Mean (Standard Deviation); unit: kg/m^2] | 32.1 (7.74) | 31.8 (7.75) | 32.0 (7.74)
Weight [Mean (Standard Deviation); unit: lbs] | 207.5 (50.99) | 206.1 (51.33) | 206.8 (51.16)
Height [Mean (Standard Deviation); unit: in] | 67.5 (3.60) | 67.5 (3.62) | 67.5 (3.61)
Donor Status [Count of Participants; unit: Participants]
  Repeat | 1608 | 1618 | 3226
  First-Time | 109 | 108 | 217
Hematocrit [Mean (Standard Deviation); unit: percentage of red blood cells] | 45.5 (3.81) | 45.4 (3.77) | 45.5 (3.79)

OUTCOME MEASURES:

1. Primary Outcome: Rate of Significant Hypotensive Adverse Events
Description: The incidence rate of at least one significant hypotensive (vasovagal/hypovolemia) adverse event according to the plasma center adverse event reporting system, based on IQPP definitions of Signs/Symptoms/Findings.
  Significant adverse events are defined as such events that fulfill the Signs/Symptoms/Findings of IQPP Donor Adverse Events (DAE) classifications 1.2 through 1.6 per the modified, symptoms-based approach following the plasma center adverse event reporting system.
  A Model Based Prediction method was used for this outcome.
Time Frame: Up to approximately 3 months (total trial duration during which donors could donate), depending on time of enrollment into the trial.
Measure: Number (95% Confidence Interval); unit: % of significant hypotensive AEs
Units Other Than Participants: Donations
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 1717 | 1726
Number analyzed (Donations) | 11362 | 11775
% of significant hypotensive AEs | .035 [.010 to .094] | .051 [.020 to .114]

2. Secondary Outcome: Rate of Severe Hypotensive Adverse Events
Description: Incidence rate of severe hypotensive (vasovagal/hypovolemia) adverse events according to the plasma center adverse event reporting system, based on the IQPP definitions of Signs/Symptoms/Findings, per donation in donors undergoing plasmapheresis.
  *Only two severe (1.5) adverse events were observed: one in the experimental group and one in the control group. As the secondary analysis for severe hypotensive adverse events was to be conducted only if there were more than 2 severe hypotensive (vasovagal/hypovolemia) adverse events in any of the two study groups, no formal statistical analysis was performed.
Time Frame: Up to approximately 3 months, depending on time of enrollment into the trial.
Measure: Number; unit: Severe Hypotensive Adverse Events
Units Other Than Participants: Donations
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 1717 | 1726
Number analyzed (Donations) | 11362 | 11775
Severe Hypotensive Adverse Events | 1 | 1

3. Secondary Outcome: Rate of Significant Hypotensive Adverse Events Relative to Volume
Description: Incidence rate of significant hypotensive (vasovagal/hypovolemia) adverse events according to the plasma center adverse event reporting system, based on the IQPP definitions of Signs/Symptoms/Findings, relative to the actual plasma volume collected.
  *The outcome is reported as the expected number of significant hypotensive adverse events per 10,000 L of collected plasma. This outcome was calculated using the total number of significant hypotensive adverse events and the total amount of plasma collected, then normalized to 10,000 L of collected plasma.
Time Frame: Up to approximately 3 months, depending on time of enrollment into the trial.
Population: This analysis was performed on the PP (per protocol) population, defined as all donations where the apheresis procedure was successfully completed collecting at least 90% of target plasma volume as well as all donations associated with a significant hypotensive (vasovagal/hypovolemia) adverse event according to the plasma center adverse event reporting system, based on the IQPP definitions of Signs/Symptoms/Findings.
Measure: Number; unit: No. of AEs per 10,000L of Plasma
Units Other Than Participants: Donations
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 1684 | 1689
Number analyzed (Donations) | 10984 | 11458
No. of AEs per 10,000L of Plasma | 4.27 | 6.65

4. Secondary Outcome: Time From Start of Collection to First Significant Hypotensive Adverse Event
Description: Time from start of plasmapheresis "Begin Draw" to the first significant hypotensive (vasovagal/hypovolemia) adverse event according to the plasma center adverse event reporting system, based on the IQPP definitions of Signs/Symptoms/Findings.
Time Frame: Up to approximately 3 months, depending on time of enrollment into the trial.
Measure: Mean (Standard Deviation); unit: minutes
Units Other Than Participants: Donations
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 1717 | 1726
Number analyzed (Donations) | 11362 | 11775
minutes | 30.41 (16.52) | 51.59 (17.09)

5. Secondary Outcome: Rate of Significant Hypotensive Adverse Events Relative to Bodyweight
Description: Incidence rate of significant hypotensive (vasovagal/hypovolemia) adverse events according to the plasma center adverse event reporting system, based on the IQPP definitions of Signs/Symptoms/Findings, in the subgroups of donors with a bodyweight of less than or equal to 130 lbs and those greater than 130 lbs.
  *Note: Due to the absence of AE in the subgroup of donors with bodyweight of ≤130 lbs, no formal statistical analysis was performed.
Time Frame: Up to approximately 3 months, depending on time of enrollment into the trial.
Population: The total number of Participants Analyzed is more than the total population of donors in the study as some donors moved from one bodyweight group to the other throughout their participation in the study. Therefore, this analysis was done at the donation level, based on the bodyweight of each donor at the time of each donation. The number of donations are therefore also listed.
Measure: Number (95% Confidence Interval); unit: % of significant hypotensive AEs
Units Other Than Participants: Donations
Groups:
- Experimental Group With Weight ≤ 130 Lbs; Experimental Group With Weight > 130 Lbs: Plasma collection using a modified version (version 1.3.90) of NexSys PCS embedded software installed on current FDA-cleared NexSys PCS device hardware (PCS-300-US), with the new plasma collection feature enabled.
  Updated Plasma Collection Feature: Plasma collection using a novel, patented system that supports a more individualized collection approach.
- Control Group With Weight ≤ 130 Lbs; Control Group With Weight > 130 Lbs: Plasma collection using a modified version (version 1.3.90) of NexSys® PCS embedded software installed on current FDA-cleared NexSy PCS device hardware (PCS-300-US), with the new plasma collection feature disabled.
  Current Plasma Collection Approach: Plasma collection using the current collection approach.
Arm/Group | Experimental Group With Weight ≤ 130 Lbs | Control Group With Weight ≤ 130 Lbs | Experimental Group With Weight > 130 Lbs | Control Group With Weight > 130 Lbs
Number analyzed (Participants) | 53 | 61 | 1671 | 1689
Number analyzed (Donations) | 251 | 287 | 11111 | 11488
% of significant hypotensive AEs | 0 [0 to 0] | 0 [0 to 0] | .036 [.010 to .096] | .052 [.020 to .117]

6. Secondary Outcome: Rate of Significant Hypotensive Adverse Events Relative to BMI
Description: Incidence rate of significant hypotensive (vasovagal/hypovolemia) adverse events according to the plasma center adverse event reporting system, based on the IQPP definitions of Signs/Symptoms/Findings, in the subgroups of donors with a body mass index (BMI) of less than or equal to 30 and of those greater than 30.
Time Frame: Up to approximately 3 months, depending on time of enrollment into the trial.
Population: The total number of Participants Analyzed is more than the total population of donors in the study as some donors moved from one BMI group to the other throughout their participation in the study. Therefore, this analysis was done at the donation level, based on the BMI of each donor at the time of each donation. The number of donations are therefore also listed.
Measure: Number (95% Confidence Interval); unit: % of significant hypotensive AEs
Units Other Than Participants: Donations
Groups:
- Experimental Group With BMI ≤ 30; Experimental Group With BMI > 30: Plasma collection using a modified version (version 1.3.90) of NexSys PCS embedded software installed on current FDA-cleared NexSys PCS device hardware (PCS-300-US), with the new plasma collection feature enabled.
  Updated Plasma Collection Feature: Plasma collection using a novel, patented system that supports a more individualized collection approach.
- Control Group With BMI ≤ 30 Lbs; Control Group With BMI > 30: Plasma collection using a modified version (version 1.3.90) of NexSys® PCS embedded software installed on current FDA-cleared NexSy PCS device hardware (PCS-300-US), with the new plasma collection feature disabled.
  Current Plasma Collection Approach: Plasma collection using the current collection approach.
Arm/Group | Experimental Group With BMI ≤ 30 | Control Group With BMI ≤ 30 Lbs | Experimental Group With BMI > 30 | Control Group With BMI > 30
Number analyzed (Participants) | 802 | 872 | 1000 | 965
Number analyzed (Donations) | 4638 | 4981 | 6724 | 6794
% of significant hypotensive AEs | .043 [.001 to .168] | .020 [-.009 to .126] | .03 [.001 to .116] | .074 [.026 to .178]

7. Secondary Outcome: Rate of Significant Hypotensive Adverse Events Relative to Donor Status
Description: Incidence rate of significant hypotensive (vasovagal/hypovolemia) adverse events according to the plasma center adverse event reporting system, based on the IQPP definitions of Signs/Symptoms/Findings, in the subgroups of donors defined by their respective status as a first-time donor or repeat donor.
Time Frame: Up to approximately 3 months, depending on time of enrollment into the trial.
Measure: Number (95% Confidence Interval); unit: % of significant hypotensive AEs
Units Other Than Participants: Donations
Groups:
- Experimental Group - First-Time Donor; Experimental Group - Repeat Donor: Plasma collection using a modified version (version 1.3.90) of NexSys PCS embedded software installed on current FDA-cleared NexSys PCS device hardware (PCS-300-US), with the new plasma collection feature enabled.
  Updated Plasma Collection Feature: Plasma collection using a novel, patented system that supports a more individualized collection approach.
- Control Group - First-Time Donor; Control Group - Repeat Donor: Plasma collection using a modified version (version 1.3.90) of NexSys® PCS embedded software installed on current FDA-cleared NexSy PCS device hardware (PCS-300-US), with the new plasma collection feature disabled.
  Current Plasma Collection Approach: Plasma collection using the current collection approach.
Arm/Group | Experimental Group - First-Time Donor | Control Group - First-Time Donor | Experimental Group - Repeat Donor | Control Group - Repeat Donor
Number analyzed (Participants) | 109 | 108 | 1608 | 1618
Number analyzed (Donations) | 419 | 405 | 10943 | 11370
% of significant hypotensive AEs | 0 [0 to 1.095] | .247 [0 to 1.531] | .037 [.011 to .098] | .044 [.016 to .106]

8. Secondary Outcome: Rate of Significant Hypotensive Adverse Events Relative to Gender
Description: Incidence rate of significant hypotensive (vasovagal/hypovolemia) adverse events according to the plasma center adverse event reporting system, based on the IQPP definitions of Signs/Symptoms/Findings, in the subgroups of donors defined by their gender.
Time Frame: Up to approximately 3 months, depending on time of enrollment into the trial.
Measure: Number (95% Confidence Interval); unit: % of significant hypotensive AEs
Units Other Than Participants: Donations
Groups:
- Experimental Group - Female Donor; Experimental Group - Male Donor: Plasma collection using a modified version (version 1.3.90) of NexSys PCS embedded software installed on current FDA-cleared NexSys PCS device hardware (PCS-300-US), with the new plasma collection feature enabled.
  Updated Plasma Collection Feature: Plasma collection using a novel, patented system that supports a more individualized collection approach.
- Control Group - Female Donor; Control Group - Male Donor: Plasma collection using a modified version (version 1.3.90) of NexSys® PCS embedded software installed on current FDA-cleared NexSy PCS device hardware (PCS-300-US), with the new plasma collection feature disabled.
  Current Plasma Collection Approach: Plasma collection using the current collection approach.
Arm/Group | Experimental Group - Female Donor | Control Group - Female Donor | Experimental Group - Male Donor | Control Group - Male Donor
Number analyzed (Participants) | 605 | 601 | 1112 | 1125
Number analyzed (Donations) | 3485 | 3739 | 7877 | 8036
% of significant hypotensive AEs | .048 [.014 to .130] | .07 [.028 to .155] | .028 [.010 to .066] | .040 [.018 to .082]

9. Secondary Outcome: Total Volume
Description: Total plasma volume collected per procedure.
Time Frame: Up to approximately 3 months, depending on time of enrollment into the trial.
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: mL
Units Other Than Participants: Donations
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 1684 | 1689
Number analyzed (Donations) | 10984 | 11458
mL | 841.69 [636 to 1000] | 777.84 [625 to 801]

ADVERSE EVENTS:
Time Frame: Adverse Events were monitored and collected for all donations of study participants throughout the entire duration of the clinical trial, approximately 3 months.
Description: For the purposes of this clinical trial, all adverse events (AEs) were defined and categorized according to established local guidelines and operating procedures and in accordance with IQPP definitions of Signs/Symptoms/Findings.
Arm/Group | Experimental Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/1717 | 0/1726
Serious Adverse Events (participants affected / at risk) | 0/1717 | 0/1726
Other Adverse Events (participants affected / at risk) | 76/1717 | 66/1726
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Group (N=1717) | Control Group (N=1726)
IQPP 9.1 Other (Nervous system disorders) | 1 (1) | 0 (0) — A reaction that does not fall into any other IQPP category. In this event, donor reported feeling dizzy during standard screening, prior to any plasmapheresis or study activities.
IQPP 8.1 Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — May include Anxiousness / Anxiety; Carpopedal Spasms; Chest Tightness; Dry Mouth; Paresthesia (Perioral -Tingling/Numbness); Paresthesia (Peripheral - Hands/Feet); Respiration, Rapid; Restlessness; Shaking; Shortness of Breath; or Tetany.
IQPP 7.1 Allergic: Local (Immune system disorders) | 3 (3) | 5 (5) — May include Itching; Rash/Hives; or Redness.
IQPP 4.2 Citrate Reaction: Moderate (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — May include Carpopedal Spasms; Chest Pressure; Cold Extremities; Chills; Muscle Tightness/Cramping; Nausea; Pallor, Pale Skin or Lips; Shortness of Breath; Sneezing/Nasal Congestion; Tetany (Transient); Tremors; Twitching; or Vomiting.
IQPP 4.1 Citrate Reaction: Minor (Injury, poisoning and procedural complications) | 2 (2) | 3 (3) — May include Metallic Taste; Paresthesia (Perioral - Lips (Tingling/Numbness); or Paresthesia (Peripheral - Hands/Feet Tingling/Numbness).
IQPP 3.3 Local Injury Related to Phlebotomy: Hematoma/Bruise (complicated) (Injury, poisoning and procedural complications) | 12 (12) | 16 (16) — May include Paresthesias, Numbness/Tingling of Fingers, Hand, or Arm; Pressure; Redness; Restricted Movement; Shooting Pain Down Arm; Significant Pain; Skin Discoloration; Swelling; Tenderness; Warmth; or Weakness of Arm.
IQPP 3.2 Local Injury Related to Phlebotomy: Hematoma/Bruise (uncomplicated) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — May include Mild Pain; No Restriction of Movement; Skin Discoloration; or Swelling.
3.1 Local Injury Related to Phlebotomy: Nerve Irritation (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) — May include Immediate Intense Pain at Site; Paresthesias, Numbness/Tingling of Fingers, Hand, or Arm; Shooting Pain Down Arm; or Weakness of Arm.
IQPP 1.5 Hypotensive (Vasovagal/Hypovolemia); Severe (With or Without LOC) (Vascular disorders) | 1 (1) | 1 (1) — This reaction may or may not include LOC and may include Chest Pain, Convulsions/Seizures, Loss of Bladder/Bowel
IQPP 1.4 Hypotensive (Vasovagal/Hypovolemia): LOC (prolonged) (Vascular disorders) | 0 (0) | 1 (1) — In this reaction, LOC lasts approximately sixty seconds or longer.
IQPP 1.3 Hypotensive: LOC (brief) (Vascular disorders) | 1 (1) | 1 (1) — In this reaction, LOC lasts approximately less than sixty seconds.
IQPP 1.2 Hypotensive: Prefaint, No LOC (Moderate): (Vascular disorders) | 2 (2) | 3 (3) — This reaction includes vomiting.
IQPP 1.1 Hypotensive: Prefaint, No LOC (Minor) (Vascular disorders) | 56 (63) | 38 (42) — May include one or more of minor symptoms, e.g., abdominal cramps, auditory disturbance, chills or shivering, clammy, cold extremities, dizziness, nausea, sweating, weakness.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site and Investigator shall not publish, disclose, present or use for instruction any Results arising out of its conduct of the Study at the Site without the express prior written consent of Sponsor, except to the extent required by applicable law. Sponsor shall have final review and approval rights for any authorized publication by Investigator, including but not limited to publication strategy, publication decisions, publication content and authorship decisions.

DOCUMENTS (2):
  • Statistical Analysis Plan (2020-04-26): https://cdn.clinicaltrials.gov/large-docs/23/NCT04320823/SAP_000.pdf
  • Study Protocol (2020-02-19): https://cdn.clinicaltrials.gov/large-docs/23/NCT04320823/Prot_001.pdf